CLINICAL TRIAL: NCT05623085
Title: Comparison of the Effects of Yoga and Aerobic Exercise Training in Primary Dysmenorrhea
Brief Title: Yoga and Aerobic Exercise Training in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA- 21091
Record Dates: First submitted 2022-10-31; First posted 2022-11-21 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Menstrual Pain; Dysmenorrhea
Keywords: Menstrual Pain; Uterine Bleeding; Yoga exercise; Aerobic exercise; Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea; Uterine Hemorrhage | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Aerobic exercise group with 8 weeks of individualized exercise according to the Karvonen protocol (heart rate reserve percentage-% HR). Exercise training will be 30 minutes at 50% of HR between weeks 0-2, 45 minutes at 50% of HR between weeks 2-4, 45 minutes at 60% of HR between weeks 4-6 and 6-8 weeks It will be done on the treadmill 3 days a week, for 60 minutes at 60% of HR between weeks. The treadmill speed will be adjusted during exercise to maintain the set target heart rate level.
  Interventions: Other: Aerobic exercise
- Yoga Exercise (Active Comparator): Yoga exercise group with 8 weeks of individualized exercise program. Exercise training will be done 3 days a week. The duration of the exercise will be adjusted to be the same as the aerobic exercise group.
  Interventions: Other: Yoga exercise

INTERVENTIONS:
Other: Aerobic exercise — Individuals in this group will be given 8-week individualized exercise according to the Karvonen protocol (heart rate reserve percentage-% HR). Exercise training will be 30 minutes at 50% of HR between weeks 0-2, 45 minutes at 50% of HR between weeks 2-4, 45 minutes at 60% of HR between weeks 4-6 and 6-8 weeks It will be done on the treadmill 3 days a week, for 60 minutes at 60% of HR between weeks. The treadmill speed will be adjusted during exercise to maintain the set target heart rate level.
  Arms: Aerobic Exercise
Other: Yoga exercise — Individuals in this group will be given 8-week individualized yoga exercise including stretching, relaxing, strength training. Exercise training will be done 3 days a week. The duration of the exercise will be adjusted to be the same as the aerobic exercise group.
  Arms: Yoga Exercise

SUMMARY:
The aim of this study is to compare the effects of aerobic exercise and yoga exercises on menstrual pain parameters (pain severity and duration, analgesic usage), uterine artery blood flow, menstrual stress level, physical fitness, anxiety/depressive symptom level, quality of life and sleep quality in individuals with primary dysmenorrhea. This study is a prospective, parallel group, randomized study. Three days a week for eight weeks, the participants in this study will receive individualized yoga and aerobic exercise.

In the literature, there are no studies comparing the effectiveness of aerobic exercise and yoga in the management of PD, which is a public health problem that seriously affects women's lives. Especially when aerobic exercise and yoga exercises are considered, there is no study on how much the features such as uterine artery blood flow and physical fitness sub-parameters have changed with these two commonly used exercise types separately in the management of PD.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of aerobic exercise and yoga exercises on menstrual pain parameters (pain severity and duration, analgesic usage), uterine artery blood flow, menstrual stress level, physical fitness, anxiety/depressive symptom level, quality of life and sleep quality in individuals with primary dysmenorrhea. This study is a prospective, parallel group, randomized study.

It was planned to enroll 44 individuals with Primary Dysmenorrhea in this randomized study. A physical therapist is responsible for all assessments.

Participants were included in one of two treatment groups (G1: Aerobic exercise; G2: Yoga exercise).

In the literature, there are no studies comparing the effectiveness of aerobic exercise and yoga in the management of PD, which is a public health problem that seriously affects women's lives. Especially when aerobic exercise and yoga exercises are considered, there is no study on how much the features such as uterine artery blood flow and physical fitness sub-parameters have changed with these two commonly used exercise types separately in the management of PD.

The results of our study show that norm values can be established by evaluating uterine arterial blood flow and physical fitness, instead of focusing on pharmacological treatment and classical nonpharmacological approaches (warm application, transcutaneous electrical nerve stimulation (TENS), acupuncture, etc.) in individuals with PD. It is aimed to develop new exercise protocols that can be done easily. It is expected that our results, which we will obtain in the light of the original values of our research, will contribute to the literature and guide future studies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who do not have any known disease (systemic, metabolic, etc.),
* No complaints of acute or chronic pain other than dysmenorrhea,
* Meeting the primary dysmenorrhea criteria outlined in the Primary Dysmenorrhea Consensus Guide (onset of menstrual pain 6-24 months after menarche, menstrual pain lasting 8-72 hours, and the most severe pain felt on the 1st or 2nd day of menstruation),
* Have a regular menstrual cycle (28± 7 days),
* The severity of menstrual pain in the last 6 months is ≥ 4 cm according to the Visual Analogue Scale,
* 18 years and over,
* Nulligravid (unborn)
* Volunteer female individuals who gave consent to participate in the study

Exclusion Criteria:

* Individuals undergoing pelvic surgery,
* Having a history and/or finding of secondary dysmenorrhea,
* Receiving alternative treatment,
* Using intrauterine contraceptive device or birth control pill,
* Individuals with situations where exercise is contraindicated (answering yes to any of the 7 questions on the exercise readiness scale),
* Not complying with the requirements of the research protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Menstrual pain severity | Change in severity of menstrual pain from baseline up to end of 8th week, 3rd month, and 6th month.
  As primary outcome measures, the highest menstrual pain severity perceived by the participants in their last menstruation and the average of the pain severity in the first 3 days of their menstruation will be evaluated. A 10-cm VAS from zero (no pain at all) to 10 (the worst pain I have ever felt) will be used to determine the severity of menstrual pain. Individuals will be asked to mark the severity of pain they felt in the first 3 days of their last menstruation on 3 separate VAS lines.

SECONDARY OUTCOMES:
Uterine artery blood flow | Change in uterine artery blood flow from baseline up to end of 8th week.
  Determination of uterine artery blood flow changes will be made with Doppler US imaging device. Uterine arterial blood flow will be determined by recording the systole / diastole ratios (S / D), pulsatility indices (PI) and resistance indices (RI) values in the first 3 days of the menstrual cycle of individuals.
Body mass index | Change in body mass index from baseline up to end of 8th week, 3rd month, and 6th month.
  Evaluation of body mass index will be done by weighing scale. Results will be presented in kg/m2.
body fat percentage | Change in body fat percentage from baseline up to end of 8th week, 3rd month, and 6th month.
  Evaluation of body fat percentage will be done by weighing scale. Results will be presented in %.
body fat amount | Change in body fat amount from baseline up to end of 8th week, 3rd month, and 6th month.
  Evaluation of body fat amount will be done by weighing scale. Results will be presented in kg.
lean body weight ratio | Change in lean body weight ratio from baseline up to end of 8th week, 3rd month, and 6th month.
  Evaluation of lean body weight ratio will be done by weighing scale. Results will be presented in %.
Lean body weight | Change in lean body weight ratio from baseline up to end of 8th week, 3rd month, and 6th month.
  Evaluation of lean body weight ratio will be done by weighing scale. Results will be presented in kg.
Cardiovascular fitness | Change in cardiovascular fitness from baseline up to end of 8th week, 3rd month, and 6th month.
  Cardiovascular fitness will be evaluated with the "6-minute walk test". For this test, which evaluates functional performance; Marking will be made at both starting points of a distance of 30 meters in the corridor. Individuals will be asked to walk for 6 minutes at the highest speed without running, and at the end of 6 minutes, the distance they walked will be recorded in meters. During the exercise test, vital signs such as blood pressure, heart rate, fatigue, shortness of breath, oxygen saturation of all individuals will be recorded before and immediately after the test.
Muscular static endurance | Change in muscular static endurance from baseline up to end of 8th week, 3rd month, and 6th month.
  For the abdominal static endurance test, a board will be used to position the patient in 60º flexion. The subjects will be positioned with the trunk at 60°, the hips and knees flexed at 90°, and the hands on the opposite shoulders, leaning against the board. The board will be pulled back 10 cm and the patient will be asked to keep his isometric position as much as possible by contracting his abdominal muscles. As soon as the subject's body touches the board, the test will be terminated and the time to hold the position will be recorded in seconds. The test is continued for a maximum of 120 seconds and after 120 seconds the test will be stopped.
Muscular dynamic endurance | Change in muscular dynamic endurance from baseline up to end of 8th week, 3rd month, and 6th month.
  30 seconds sit-up test will be used for dynamic endurance. In the 30-second sit-up test, individuals will be asked to stand up to the level of the lower angle of the scapula and return to the starting position, with the knees flexed at 90 degrees, the hands on the back of the neck and the soles of the feet on the ground, with the command to start in the supine position to evaluate the dynamic endurance of the abdominal muscles. The exact and correct number of starts during 30 seconds will be recorded as the test score.
Muscle strength (for lower extremity) | Change in muscular strength from baseline up to end of 8th week, 3rd month, and 6th month.
  Dominant side knee extension strength for the lower extremity will be measured with the Nicholas Manual Muscle Tester.
Muscle strength (for upper extremity) | Change in muscular strength from baseline up to end of 8th week, 3rd month, and 6th month.
  For upper extremity muscle strength, the grip strength of the dominant hand will be measured with a Hand grip dynamometer.
Flexibility | Change in flexibility from baseline up to end of 8th week, 3rd month, and 6th month.
  It will be evaluated with the sit-reach test. Individuals will be asked to perform maximum trunk flexion with both hands on top of each other in a long sitting position with legs straight. The distance between the tip of the hand and the board against the soles of the feet will be measured. The distance will be recorded in +/- centimeters (cm).
Menstrual stress level | Change in menstrual stress level from baseline up to end of 8th week, 3rd month, and 6th month.
  The complaints of individuals in the menstrual, premenstrual and intermenstrual periods will be evaluated in the Menstrual Distress Complaint List.
Anxiety/depressive symptom level | Change in anxiety/depressive symptom level from baseline up to end of 8th week, 3rd month, and 6th month.
  Anxiety and depressive symptom levels of individuals will be evaluated with the Depression Anxiety Stress Scale.
Quality of life level | Change in quality of life level from baseline up to end of 8th week, 3rd month, and 6th month.
  The quality of life of individuals will be evaluated with the World Health Organization Quality of Life Scale-Short Form. In the scale consisting of 5 subsections, each section score varies between 4 and 20. Higher scores indicate higher quality of life.
Sleep quality | Change in sleep quality level from baseline up to end of 8th week, 3rd month, and 6th month.
  Sleep quality of individuals will be evaluated with the Women's Health Initiative Insomnia Scale. The higher the score, the higher the degree of insomnia.
Perception of improvement | Change in perception of improvement from baseline up to end of 8th week, 3rd month, and 6th month..
  A 3-point Likert-type scale will be used to evaluate the subjective perception of improvement of individuals. An increase in the score indicates that the perception of improvement increases.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Özgül, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Gamze Nalan Çinar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wickstrom K, Edelstam G. Minimal clinically important difference for pain on the VAS scale and the relation to quality of life in women with endometriosis. Sex Reprod Healthc. 2017 Oct;13:35-40. doi: 10.1016/j.srhc.2017.05.004. Epub 2017 May 25. PMID 28844356
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Guimaraes AC, Vaz MA, De Campos MI, Marantes R. The contribution of the rectus abdominis and rectus femoris in twelve selected abdominal exercises. An electromyographic study. J Sports Med Phys Fitness. 1991 Jun;31(2):222-30. PMID 1836517
- [Background] Bianco A, Lupo C, Alesi M, Spina S, Raccuglia M, Thomas E, Paoli A, Palma A. The sit up test to exhaustion as a test for muscular endurance evaluation. Springerplus. 2015 Jul 2;4:309. doi: 10.1186/s40064-015-1023-6. eCollection 2015. PMID 26155448
- [Background] Arnold CM, Warkentin KD, Chilibeck PD, Magnus CR. The reliability and validity of handheld dynamometry for the measurement of lower-extremity muscle strength in older adults. J Strength Cond Res. 2010 Mar;24(3):815-24. doi: 10.1519/JSC.0b013e3181aa36b8. PMID 19661831
- [Background] Moos RH. The development of a menstrual distress questionnaire. Psychosom Med. 1968 Nov-Dec;30(6):853-67. doi: 10.1097/00006842-196811000-00006. No abstract available. PMID 5749738
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Levine DW, Kripke DF, Kaplan RM, Lewis MA, Naughton MJ, Bowen DJ, Shumaker SA. Reliability and validity of the Women's Health Initiative Insomnia Rating Scale. Psychol Assess. 2003 Jun;15(2):137-48. doi: 10.1037/1040-3590.15.2.137. PMID 12847774
- [Background] Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989 Dec;10(4):407-15. doi: 10.1016/0197-2456(89)90005-6. PMID 2691207